CLINICAL TRIAL: NCT01709149
Title: A Phase IIb, Multi-National, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of CK-2017357 in Patients With Amyotrophic Lateral Sclerosis (ALS) (BENEFIT-ALS)
Brief Title: Study of Safety, Tolerability & Efficacy of CK-2017357 in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 4026
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — CK-2017357; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CK-2017357 (Experimental): 125 mg tablets
  Interventions: Drug: CK-2017357; Drug: Riluzole
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Other: Placebo tablets; Drug: Riluzole

INTERVENTIONS:
Drug: CK-2017357 — CK-2017357 125 mg tablets twice daily
  Other Names: tirasemtiv
  Arms: CK-2017357
Other: Placebo tablets — Tablets
  Arms: Placebo
Drug: Riluzole — Tablets
  Other Names: Rilutek

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of CK-2017357 when taken with or without riluzole (also called Rilutek®) in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
The length of the study, including screening, dosing, and follow-up, is approximately 20 weeks. After a one-week open-label phase during which all patients will receive CK-2017357 125 milligrams (mg) twice daily, patients who tolerate the open-label 125 mg of CK-2017357 will be randomized one to one (fifty-fifty) to receive double-blind CK-2017357 or matching placebo. The CK-2017357/placebo dose will be increased no faster than weekly to each patient's highest tolerated daily dose, with a maximum of 250 mg twice daily. The dose may be decreased based on tolerability. Patients will continue treatment at the highest tolerated dose to complete a total of 12 weeks of double-blind treatment. Patients may be on riluzole or not on riluzole at study entry. Patients not on riluzole must stay off riluzole. Patients on riluzole who are getting double-blind CK-2017357 will be given riluzole at half the labeled dosage (50 mg once a day instead of 50 mg twice a day). Blood tests for safety will be performed. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF)
2. Male or female 18 years of age or older
3. A diagnosis of familial or sporadic ALS (defined as meeting the possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the World Federation of Neurology El Escorial criteria)
4. Upright Slow Vital Capacity (SVC) >50 % of predicted for age, height and sex
5. At least 4 of the 12 ALSFRS-R questions must be scored 2 or 3
6. Diminished but measurable maximum voluntary grip strength in at least one hand; i.e., between 10 and 50 pounds (females) and 10 and 70 pounds (males)
7. Able to swallow tablets without crushing
8. A caregiver (if one is needed) who can and will observe and report the patient's status
9. Pre-study clinical laboratory findings within normal range or, if outside of the normal range, deemed not clinically significant by the Investigator
10. Male patients must agree for the duration of the study and 10 weeks after the end of the study to use a condom during sexual intercourse with female partners who are of reproductive potential and to have female partners use an additional effective means of contraception (e.g., diaphragm plus spermicide, or oral contraceptives) or the male patient must agree to abstain from sexual intercourse during and for 10 weeks after the end of the study
11. Female patients must be post-menopausal (≥ 1 year) or sterilized, or, if of childbearing potential, not be breastfeeding, have a negative pregnancy test, have no intention to become pregnant during the course of the study, and use contraceptive drugs or devices as detailed in item 10 for the duration of the study and for 10 weeks after the end of the study
12. Patients must be either on a stable dose of riluzole 50 mg twice daily for at least 30 days prior to screening or have not taken riluzole for at least 30 days prior to screening and are willing not to begin riluzole use during the conduct of this study.

Exclusion Criteria:

1. Any use of non-invasive positive pressure ventilation (NIPPV, e.g. continuous positive airway pressure [CPAP] or bilevel positive airway pressure [BiPAP]) for any portion of the day, or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation
2. Patients with a diaphragm pacing system (DPS) at study entry or who anticipate DPS placement during the course of the study
3. Body Mass Index (BMI) of 19.0 kg/m2 or lower
4. Unwilling to discontinue tizanidine and theophylline-containing medications during study participation
5. Serum chloride < 100 mmol/L
6. Neurological impairment due to a condition other than ALS, including history of transient ischemic attack (TIA) within the past year
7. Presence at screening of any medically significant cardiac, pulmonary, gastrointestinal (GI), musculoskeletal, or psychiatric illness that might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety or efficacy data
8. Has taken any investigational study drug within 30 days or 5 half-lives of the prior agent, whichever is greater, prior to dosing
9. Previously received CK-2017357 in any previous clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinsy Andrews, MD, Study Director — Cytokinetics, Inc.; Jeremy Shefner, MD, PhD, Study Chair — State University of New York - Upstate Medical University; Jeremy Shefner, MD, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (75):
- United States (44):
  - Barrow Neurology, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - UC Irvine ALS & Neuromuscular Center, Orange, California
  - Coordinated Clinical Research, San Diego, California
  - California Pacific Medical Center Forbes Norris MDA/ALS Research Center, San Francisco, California
  - Hospital for Special Care, New Britain, Connecticut
  - The George Washington University, Washington D.C., District of Columbia
  - Mayo Clinic Florida Department of Neurology, Jacksonville, Florida
  - Emory University, School of Medicine, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Indiana University Department of Neurology, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St Mary's Healthcare, Grand Rapids, Michigan
  - Hennepin County Medical Center - Berman Center for Research, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Neurology Associates, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hospital for Special Surgery, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center Department of Neurology, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University, School of Medicine, Winston-Salem, North Carolina
  - Ohio State University Department of Neurology, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey Neuroscience Clinics, Hershey, Pennsylvania
  - Drexel Neurology, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - UTHSCSA Department of Neurology, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University Department of Neurology, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (12):
  - Heritage Medical Research, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - Queen's University : Kingston General, Kingston, Ontario
  - London Health Sciences, London, Ontario
  - Univ. of Toronto - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital Notre Dame (CHUM) Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Montreal Neurological Institute, Montreal, Quebec
  - CHU de Quebec: Hopital l'Enfant-Jesus, Québec, Quebec
- France (7):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpital La Timone Adulte, Marseille
  - CHU Montepellier, Montpellier
  - Hôpital Archet 1, Nice
  - Hôpital de la Salpêtrière, Paris
  - Hôpital Bretonneau, Tours
- Germany (3):
  - Charite Universitätsmedizin, Berlin
  - Hannover Medical School, Hanover
  - University of Ulm, Ulm
- Trinity College, Beaumont Hospital, Dublin, Ireland
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Carlos III, Madrid, Spain
- United Kingdom (6):
  - Barts and the London MND & the Centre Royal London Hospital, Whitechapel, London
  - Walton Centre for Neurology and Neurosurgery, Liverpool
  - Kings College Hospital NHS Foundation Trust, London
  - John Radcliffe Hospital, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth
  - Sheffield Institute for Translational Neuroscience, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with familial or sporadic amyotrophic lateral sclerosis were enrolled at 73 sites in Canada, France, Germany, Ireland, Netherlands, Spain, the United Kingdom, and the United States. The first patient was screened on 23 October 2012 and the last subject completed follow-up on 21 March 2014.
Pre-assignment Details: A total of 711 patients were enrolled in the study and began treatment with open-label tirasemtiv during the 7-day lead-in phase of the study. Patients who completed this phase were randomized (1:1) to receive either placebo (N=295) or tirasemtiv (N=301) in the double-blind treatment period.
Groups:
- Open-label lead-in Treatment: Tirasemtiv: Tirasemtiv 125 mg oral capsules administered twice daily for 7 days prior to randomization to the Double-blind treatment period.
- Double-blind Treatment: Placebo: Placebo oral capsules administered twice daily for a total of 12 weeks of double-blind dosing.
- Double-blind Treatment: Tirasemtiv: Tirasemtiv 125 mg oral capsules administered twice daily. Minimum dose was 125 mg bid and patients were up- or down-titrated over 3 to 4 weeks to the patient's maximum tolerated dose (MTD) to a maximum of 250 mg twice daily. Patients then remained at their MTD for an additional 9 weeks, for a total of 12 weeks of double-blind dosing.
Period: Open-label Lead-in Phase
Arm/Group | Open-label lead-in Treatment: Tirasemtiv | Double-blind Treatment: Placebo | Double-blind Treatment: Tirasemtiv
Started | 711 | 0 | 0
Completed | 596 | 0 | 0
Not Completed | 115 | 0 | 0
Not completed — Adverse Event | 109 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Period: Double-blind, Placebo-controlled Phase
Arm/Group | Open-label lead-in Treatment: Tirasemtiv | Double-blind Treatment: Placebo | Double-blind Treatment: Tirasemtiv
Started | 0 | 295 | 301
Completed | 0 | 269 | 204
Not Completed | 0 | 26 | 97
Not completed — Adverse Event | 0 | 12 | 78
Not completed — Withdrawal by Subject | 0 | 7 | 12
Not completed — Physician Decision | 0 | 2 | 5
Not completed — Death | 0 | 2 | 0
Not completed — not defined | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (all patients who received any study drug)
Groups:
- Did Not Complete Open-label Lead-in Treatment: Tirasemtiv 125 mg oral capsules administered twice daily for 7 days. This group started open-label treatment but discontinued early and did not receive double-blind treatment.
- Double-blind Treatment: Tirasemtiv: Tirasemtiv 125 mg oral capsules administered twice daily, which was up- or down-titrated over 3 to 4 weeks to the patient's maximum tolerated dose (MTD) to a maximum of 250 mg twice daily. Patients then remained at their MTD for an additional 9 weeks, for a total of 12 weeks of double-blind dosing.
- Total: Total of all reporting groups
Arm/Group | Did Not Complete Open-label Lead-in Treatment | Double-blind Treatment: Placebo | Double-blind Treatment: Tirasemtiv | Total
Number analyzed (Participants) | 115 | 295 | 301 | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.83) | 56.9 (11.10) | 57.0 (11.17) | 57.5 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 88 | 86 | 226
  Male | 63 | 207 | 215 | 485
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 8 | 9 | 20
  White | 102 | 250 | 259 | 611
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 34 | 26 | 68
Time since ALS symptom onset [Median (Full Range); unit: months] | 24.0 [4 to 278] | 21.0 [4 to 224] | 23.0 [5 to 272] | 22.0 [4 to 278]
Site of symptom onset [Count of Participants; unit: Participants]
  Lower limb | 43 | 110 | 116 | 269
  Upper limb | 51 | 145 | 149 | 345
  Bulbar | 20 | 40 | 35 | 95
  Respiratory | 1 | 0 | 1 | 2
El Escorial Diagnostic Criteria for ALS [Count of Participants; unit: Participants] — Per El Escorial criteria, ALS was diagnosed as: Possible (upper motor neuron [UMN] and lower motor neuron [LMN] signs in 1 region, or UMN signs in at least 2 regions, or UMN and LMN signs in 2 regions with no UMN signs rostral to LMN signs); Probable, Laboratory Supported (UMN signs in 1 or more regions and LMN signs defined by electromyography in at least 2 regions); Probable (UMN and LMN signs in 2 regions with some UMN signs rostral to the LMN signs); and Definite (UMN and LMN signs in 3 regions).
  The El Escorial criteria do not relate to grading of ALS nor to outcome.
  Participants
    Possible | 9 | 28 | 31 | 68
    Probable, laboratory supported | 15 | 57 | 63 | 135
    Probable | 46 | 119 | 103 | 268
    Definite | 45 | 91 | 104 | 240

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in ALS Functional Rating Scale-Revised (ALSFRS-R) Total Score to the Average of Values Obtained at the End of Weeks 8 and 12 of Double-blind Treatment
Description: The ALSFRS-R is used to measure the progression and severity of disease; it consists of 12 questions, assessing a patient's capability and independence in functional activities relevant to ALS, categorized in 4 domains: gross motor tasks, fine motor tasks, bulbar functions, and respiratory function. Each question is scored from 0 (indicating incapable or dependent) to 4 (normal). The total score ranges from 0 to 48, with higher scores reflecting more normal function and lower scores reflecting more impaired function.
Time Frame: Baseline, 8 weeks, 12 weeks
Population: Modified Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo oral capsules administered twice daily for a total of 12 weeks of double-blind dosing.
- Tirasemtiv: Tirasemtiv 125 mg oral capsules administered twice daily, which was up- or down-titrated over 3 to 4 weeks to the patient's maximum tolerated dose (MTD) to a maximum of 250 mg twice daily. Patients then remained at their MTD for an additional 9 weeks, for a total of 12 weeks of double-blind dosing.
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
units on a scale | -2.40 (0.246) | -2.98 (0.277)
Statistical Analysis 1: Comparison: Placebo vs Tirasemtiv; Test type: Superiority; p = 0.1140, Repeated-measures mixed model; Least squares mean difference = -0.58, 95% CI 2-sided [-1.30 to 0.14], Standard Error of Mean 0.366 — Least squares mean difference: tirasemtiv minus placebo

2. Secondary Outcome: Change From Baseline in Maximum Voluntary Ventilation (MVV) to the Average of Values Obtained at the End of Weeks 8 and 12 of Double-blind Treatment
Description: MVV was measured as the volume (in liters) of air that could be exhaled during 12 seconds of rapid deep breathing; for analysis purposes, the measured volume was extrapolated to 1 minute (to give units of L/min).
Time Frame: Baseline, 8 weeks, 12 weeks
Population: Modified Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
L/min | -4.27 (1.332) | -3.79 (1.497)
Statistical Analysis 1: Comparison: Placebo vs Tirasemtiv; Test type: Superiority; p = 0.8083, Repeated-measures mixed model; Least squares mean difference = 0.48, 95% CI 2-sided [-3.38 to 4.34], Standard Error of Mean 1.963 — Least squares mean difference: tirasemtiv minus placebo

3. Secondary Outcome: Change From Baseline in Sniff Nasal Inspiratory Pressure (SNIP) to the Average of Values Obtained at the End of Weeks 8 and 12 of Double-blind Treatment
Description: SNIP was measured at functional residual capacity, the bottom of the tidal breathing cycle, through 1 plugged nostril while the other remained open. Inspiratory pressure is a negative number where a larger negative number represents . . . A forceful, maximal inspiratory sniff was performed and a peak pressure value reported. The best result (ie, the highest number) from 5 tests was recorded as the SNIP.
Time Frame: Baseline, 8 weeks, 12 weeks
Population: Modified Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: cm H2O
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
cm H2O | -0.89 (1.103) | -4.29 (1.243)
Statistical Analysis 1: Comparison: Placebo vs Tirasemtiv; Test type: Superiority; p = 0.0372, Repeated-measures mixed model; Least squares mean difference = -3.40, 95% CI 2-sided [-6.60 to -0.20], Standard Error of Mean 1.627 — Least squares mean difference: tirasemtiv minus placebo

4. Secondary Outcome: Change From Baseline in Slow Vital Capacity (SVC) to the Average of Values Obtained at the End of Weeks 8 and 12 of Double-blind Treatment
Description: SVC was measured using a spirometer (in units of liters). Following 3 to 5 breaths at rest, the patients were instructed to take as deep an inspiration as possible followed by a maximum exhalation (blowing out all the air in their lungs). Values obtained were converted to % predicted values (ie, the test result as a percent of predicted values for the patients of similar demographic and baseline characteristics [eg, height, age, sex]).
Time Frame: Baseline, 8 weeks, 12 weeks
Population: Modified Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: % predicted
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
% predicted | -7.24 (0.691) | -2.98 (0.780)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Repeated-measures mixed model; Least squares mean difference = 4.25, 95% CI 2-sided [2.23 to 6.28], Standard Error of Mean 1.030 — Least squares mean difference: tirasemtiv minus placebo

5. Secondary Outcome: Change From Baseline in Maximum Handgrip Strength in the Weaker Hand to the Average of Values Obtained at the End of Weeks 8 and 12 of Double-blind Treatment
Description: Maximum handgrip strength was measured using an electronic hand dynamometer; patients were asked to squeeze the device with the maximum possible force.
Time Frame: Baseline, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: pounds
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
pounds | -3.54 (0.640) | -2.78 (0.714)
Statistical Analysis 1: Comparison: Placebo vs Tirasemtiv; Test type: Superiority; p = 0.4328, Repeated-measures mixed model; Least squares mean difference = 0.75, 95% CI 2-sided [-1.13 to 2.63], Standard Error of Mean 0.956 — Least squares mean difference: tirasemtiv minus placebo

6. Secondary Outcome: Change From Baseline in Handgrip Fatigability (at 60% of Target in the Weaker Hand) to the Average of Values Obtained at the End of Weeks 8 and 12 of Double-blind Treatment
Description: Handgrip fatigability was measured immediately following determination of maximum handgrip strength (via an electronic hand dynamometer). Once maximum handgrip strength was achieved, the force of the grip was timed for 2 minutes or until the grip strength had dropped to 60% of the maximum, whichever came first.
Time Frame: Baseline, 8 weeks, 12 weeks
Population: Modified Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
seconds | 1.76 (2.863) | 2.01 (3.331)
Statistical Analysis 1: Comparison: Placebo vs Tirasemtiv; Test type: Superiority; p = 0.9546, Repeated-measures mixed model; Least squares mean difference = 0.25, 95% CI 2-sided [-8.40 to 8.90], Standard Error of Mean 4.399 — Least squares mean difference: tirasemtiv minus placebo

7. Secondary Outcome: Change From Baseline in Muscle Strength Mega-Score Based on Percent Change in Muscle Strength Measurements to the Average at the End of Weeks 8 and 12 of Double-blind Treatment
Description: A hand-held dynamometer (HHD), with a scale of 0 to 300 pounds, was used to measure muscle strength and handgrip strength (bilateral); the muscle groups tested were: elbow flexion (bilateral), wrist extension (bilateral), knee extension (bilateral), and ankle dorsiflexion (bilateral). For each assessment time point, the percent change from baseline was calculated for each muscle group and handgrip strength. The muscle strength mega-score was calculated as the average of the changes (ie, percent change from baseline) observed for each muscle groups as well as handgrip strength. For this endpoint, negative values indicate a decline in muscle strength.
Time Frame: Baseline, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Tirasemtiv
Number analyzed (Participants) | 210 | 178
percent change | -10.71 (2.108) | -9.10 (2.425)
Statistical Analysis 1: Comparison: Placebo vs Tirasemtiv; Test type: Superiority; p = 0.6166, Repeated-measures mixed model; Least squares mean difference = 1.61, 95% CI 2-sided [-4.70 to 7.91], Standard Error of Mean 3.207 — Least squares mean difference: tirasemtiv minus placebo

ADVERSE EVENTS:
Time Frame: AEs were collected from the first dose of open-label study drug through 30 days after the last dose of study drug or Week 16, whichever was earlier.
Description: An AE was treatment-emergent if it started or worsened in severity after the first dose of study drug (in either the open-label or double-blind periods). For the double-blind period, if the AE started in the open-label period and continued into the double-blind period for more than 96 hours, it was assigned an onset of 96 hours after the first dose of double-blind study drug.
Arm/Group | Open-label lead-in Treatment: Tirasemtiv | Double-blind Treatment: Placebo | Double-blind Treatment: Tirasemtiv
All-Cause Mortality (participants affected / at risk) | 2/711 | 3/295 | 2/301
Serious Adverse Events (participants affected / at risk) | 13/711 | 16/295 | 27/301
Other Adverse Events (participants affected / at risk) | 525/711 | 258/295 | 291/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label lead-in Treatment: Tirasemtiv (N=711) | Double-blind Treatment: Placebo (N=295) | Double-blind Treatment: Tirasemtiv (N=301)
Confusional state (Psychiatric disorders) | 2 | 0 | 2
Depression (Psychiatric disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1
Paresis (Nervous system disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal haematoma (Nervous system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label lead-in Treatment: Tirasemtiv (N=711) | Double-blind Treatment: Placebo (N=295) | Double-blind Treatment: Tirasemtiv (N=301)
Dizziness (Nervous system disorders) | 291 | 58 | 153
Fatigue (General disorders) | 111 | 42 | 100
Nausea (Gastrointestinal disorders) | 77 | 23 | 66
Headache (Nervous system disorders) | 30 | 33 | 54
Asthenia (General disorders) | 40 | 37 | 48
Muscle spasms (Musculoskeletal and connective tissue disorders) | 30 | 16 | 45
Somnolence (Nervous system disorders) | 50 | 11 | 39
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 20 | 34
Confusional state (Psychiatric disorders) | 18 | 3 | 33
Insomnia (Psychiatric disorders) | 16 | 12 | 31
Decreased appetite (Metabolism and nutrition disorders) | 23 | 9 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 25
Dysarthria (Nervous system disorders) | 13 | 7 | 23
Contusion (Injury, poisoning and procedural complications) | 6 | 25 | 22
Diarrhoea (Gastrointestinal disorders) | 10 | 17 | 22
Anxiety (Psychiatric disorders) | 15 | 13 | 20
Nasopharyngitis (Infections and infestations) | 7 | 19 | 19
Constipation (Gastrointestinal disorders) | 11 | 17 | 19
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 17 | 19
Oedema peripheral (General disorders) | 5 | 17 | 18
Laceration (Injury, poisoning and procedural complications) | 6 | 11 | 18
Excoriation (Injury, poisoning and procedural complications) | 2 | 15 | 17
Urinary tract infection (Infections and infestations) | 5 | 14 | 17
Tremor (Nervous system disorders) | 8 | 7 | 17
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 17
Depression (Psychiatric disorders) | 8 | 10 | 16
Dysphagia (Gastrointestinal disorders) | 6 | 10 | 16
Muscle contractions involuntary (Nervous system disorders) | 15 | 8 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 20 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 12 | 15
Balance disorder (Nervous system disorders) | 10 | 3 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 17 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 17 | 9
Upper respiratory tract infection (Infections and infestations) | 3 | 15 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No